CLINICAL TRIAL: NCT04570813
Title: Art'Health: Effects of Artistic and Participative Workshops at the MAMAC of Nice on the Health of Seniors
Acronym: Art'Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-PP-21
Record Dates: First submitted 2020-09-22; First posted 2020-09-30 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Well Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artistic activities (Experimental): participants will do a 3-month cycle of weekly "artistic activities" at the MAMAC Museum," which are structured 2-h-long art-based workshops
  Interventions: Other: Artistic activies
- No artistic activities (No Intervention): The control group is composed of participants who do not take part in art-based activities,

INTERVENTIONS:
Other: Artistic activies — 12 workshops of artictic activities during 12 weeks
  Arms: artistic activities

SUMMARY:
Study with two arms, one of which receives an intervention in the form of participative artistic workshops at the MAMAC and the other was assigned as the control group. Well-being, Quality of life, Health, Apathy and Olfactory identification scales are proposed before the intervention, during the intervention at the end of each month (M1, M2, M3), 6 months after the end of the intervention (M9) and 12 months after the end of the intervention (M15).

ELIGIBILITY:
Inclusion Criteria:

1. Be 65 years of age at the time of signing the consent,
2. Having internet access and an electronic tool (smartphone and/or tablet) at home as repeated assessments will be proposed on a dedicated and secure internet platform,
3. To master the French language,
4. To be available during participatory workshop sessions at MAMAC.
5. Be affiliated to Social Security

Exclusion Criteria:

1. Do not master the French language,
2. Severe sensory and/or cognitive impairment identified by the IP and their representatives during the inclusion interview,
3. Person under guardianship, curatorship or safeguarding of justice,
4. Person unable to give or sign consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 127 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
changes of well being level | before the intervention, during the intervention at the end of each month (Month1, Month 2, Month 3), 6 months after the end of the intervention (Month 9) and 12 months after the end of the intervention (Month 15)
  well being scale assessment Warwick-Edimbourg Mental Well-Being State (WEMWBS)
  maximum value : 70 (better outcome) minimum value :14 (worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Auriane GROS, Principal Investigator — Research and Resources Memory Centre, Nice University Hospital, Nice, France
Locations (1):
- Centre Mémoire de Ressources et de Recherche, CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Payne M, Galery K, Plonka A, Lemaire J, Derreumaux A, Fabre R, Mouton A, Sacco G, Guerin O, Manera V, Robert P, Beauchet O, Gros A. Productive art engagement in a hybrid format: effects on emotions of older adults during COVID-19 pandemic. Front Public Health. 2024 Jan 26;12:1257411. doi: 10.3389/fpubh.2024.1257411. eCollection 2024. PMID 38344232